CLINICAL TRIAL: NCT02081183
Title: A Study to Evaluate the Efficacy of CellCept, Administered in a Sequential Treatment Scheme, in Delaying Progressive Renal Damage in Patients With Lupus Nephritis
Brief Title: A Study to Evaluate Efficacy of CellCept (Mycophenolate Mofetil) in Patients With Lupus Nephritis
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML18989
Record Dates: First submitted 2014-03-05; First posted 2014-03-07 (Estimated); Results first posted 2014-07-17 (Estimated); Last update posted 2014-07-17 (Estimated); Status verified 2014-06

CONDITIONS: Lupus Nephritis
MeSH Terms: conditions — Lupus Nephritis | interventions — Mycophenolic Acid; Cyclophosphamide; Prednisone

ARMS (2):
- MMF, Prednisone (Experimental): Induction Phase (Months 1 through 6): Participants received cyclophosphamide, 0.5 to (-) 1 grams per square meter (g/m^2), intravenously (IV) pulse once per month. Participants also received prednisone, 1 milligram per kilogram per day (mg/kg/day), orally (PO); the dose was reduced by 5 mg/day to a final dose of 10 mg/day.
  Maintenance Phase (Months 7 through 12): Participants received mycophenolate mofetil (MMF), 1 g/day, PO, twice daily (BID) for 2 weeks; 1.5 g/day, PO, three times daily (TID) for the next 2 weeks; 2 g/day, PO, BID for the remainder of the Maintenance Phase. Participants also received prednisone, as in the Induction Phase.
  Interventions: Drug: Mycophenolate mofetil (MMF); Drug: Cyclophosphamide, Induction Phase; Drug: Prednisone
- Maintenance Cyclophosphamide, Prednisone (Active Comparator): Induction Phase (Months 1 through 6): Participants received cyclophosphamide, 0.5 - 1 g/m^2, IV, pulse once per month. Participants also received prednisone, 1 mg/kg/day), PO; the dose was reduced by 5 mg/day to a final dose of 10 mg/day.
  Maintenance Phase (Months 7 through 12): Participants received cyclophosphamide, 0.5-1 g/m^2, IV, pulse once every 3 months. Participants also received prednisone, as in the Induction Phase.
  Interventions: Drug: Cyclophosphamide, Maintenance Phase; Drug: Cyclophosphamide, Induction Phase; Drug: Prednisone

INTERVENTIONS:
Drug: Mycophenolate mofetil (MMF) — 1 g/day, PO BID for 2 weeks; 1.5 g/day PO TID for the next 2 weeks; and 2 g/day PO BID for the remainder of the Maintenance Phase.
  Other Names: CellCept
  Arms: MMF, Prednisone
Drug: Cyclophosphamide, Maintenance Phase — 0.5-1 g/m^2 IV pulse once every 3 months
  Arms: Maintenance Cyclophosphamide, Prednisone
Drug: Cyclophosphamide, Induction Phase — 0.5 - 1 g/m^2 IV pulse once per month
Drug: Prednisone — 1 mg/kg PO once per day; reduced by 5 mg every 2 weeks up to 20 mg/day; followed by a reduction of 2.5 mg every 2 weeks until reaching the maintenance phase of 10 mg/day.

SUMMARY:
This study will compare the efficacy of CellCept [0.5-2 grams per day (g/day) orally (p.o.)] and cyclophosphamide [0.5-1 grams per square meter (g/m2) quarterly] as maintenance treatment for patients with lupus nephritis. All patients will receive induction treatment with cyclophosphamide (0.5-1g/m2 monthly) for 6 months, and will then be randomized to the maintenance phase of the study for a further 6 months, followed by 6 months of treatment-free follow-up. The anticipated time on study treatment is 12 months.

ELIGIBILITY:
Inclusion Criteria:

* adult patients >=18 years of age;
* diagnosis of systemic lupus erythematosus and lupus nephritis (class III, IV or V).

Exclusion Criteria:

* patients who have received cytotoxic drugs in previous 8 weeks;
* systemic infections;
* hepatitis B or C, or HIV.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2006-03; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (2):
- Venezuela (2):
  - Barquisimeto
  - Caracas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Protocol Approved by National Regulatory Agency on 25 October 2005 and inclusion period ended on 21 January 2008, on three investigational sites but only two sites included patients. Sites were selected in public health care systems.
Pre-assignment Details: Screening period include only the assessments to verified the inclusion and exclusion criteria's from ICF signature until base line visit (first dose day), no washout or run in period was expected.
Groups:
- Mycophenolate Mofetil (MMF), Prednisone: Induction Phase (Months 1 through 6): Participants received cyclophosphamide, 0.5 to (-) 1 grams per square meter (g/m^2), intravenously (IV) once per month. Participants also received prednisone, 1 milligram per kilogram per day (mg/kg/day), tablets (or methylprednisolone IV), orally (PO); the dose was reduced by 5 mg every 2 weeks up to 20 mg/day, then reduced by 2.5 mg every 2 weeks to a final maintenance dose of 10 mg/day.
  Maintenance Phase (Months 7 through 12): Participants received MMF, 500 mg, tablets or capsules, PO, twice daily (BID) for 2 weeks; 500 mg, PO, three times daily (TID) for the next 2 weeks; 1 g, PO, BID for the remainder of the Maintenance Phase. Participants continued to receive maintenance prednisone (10 mg/day), as in the Induction Phase.
- Cyclophosphamide, Prednisone: Induction Phase (Months 1 through 6): Participants received cyclophosphamide, 0.5 -1 g/m^2, IV once per month. Participants also received prednisone, 1 mg/kg/day, tablets (or methylprednisolone IV), PO; the dose was reduced by 5 mg every 2 weeks up to 20 mg/day, then reduced by 2.5 mg every 2 weeks to a final maintenance dose of 10 mg/day.
  Maintenance Phase (Months 7 through 12): Participants received cyclophosphamide, 0.5-1 g/m^2, IV, once every 3 months. Participants continued to receive maintenance prednisone (10 mg/day), as in the Induction Phase.
Period: Overall Study
Arm/Group | Mycophenolate Mofetil (MMF), Prednisone | Cyclophosphamide, Prednisone
Started | 5 | 6
Completed | 1 | 2
Not Completed | 4 | 4
Not completed — Lost to Follow-up | 0 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Other | 3 | 3

BASELINE CHARACTERISTICS:
Population: No baseline analysis was performed because the study was terminated early.
Groups:
- MMF, Prednisone: Induction Phase (Months 1 through 6): Participants received cyclophosphamide, 0.5 -1 g/m^2, IV once per month. Participants also received prednisone, 1 mg/kg/day, tablets (or methylprednisolone IV), PO; the dose was reduced by 5 mg every 2 weeks up to 20 mg/day, then reduced by 2.5 mg every 2 weeks to a final maintenance dose of 10 mg/day.
  Maintenance Phase (Months 7 through 12): Participants received MMF, 500 mg, tablets or capsules, PO, twice daily (BID) for 2 weeks; 500 mg, PO, three times daily (TID) for the next 2 weeks; 1 g, PO, BID for the remainder of the Maintenance Phase. Participants continued to receive maintenance prednisone (10 mg/day), as in the Induction Phase.
- Cyclophosphamide, Prednisone: Induction Phase (Months 1 through 6): Participants received cyclophosphamide, 0.5 -1 g/m^2, IV once per month. Participants also received prednisone, 1 mg/kg/day, tablets (or methylprednisolone IV) PO; the dose was reduced by 5 mg every 2 weeks up to 20 mg/day, then reduced by 2.5 mg every 2 weeks to a final maintenance dose of 10 mg/day.
  Maintenance Phase (Months 7 through 12): Participants received cyclophosphamide, 0.5-1 g/m^2, IV, once every 3 months. Participants continued to receive maintenance prednisone (10 mg/day), as in the Induction Phase.
- Total: Total of all reporting groups
Arm/Group | MMF, Prednisone | Cyclophosphamide, Prednisone | Total
Number analyzed (Participants) | 5 | 6 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 6 | 11
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 10
  Male | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Venezuela | 5 | 6 | 11

OUTCOME MEASURES:

1. Primary Outcome: Creatinine Clearance
Description: Creatinine clearance in an indicator of kidney function. An increased level of creatinine in the blood indicates decreased kidney function. Normal adult values are 97 to 137 milliliters per minute (mL/min) for males and 88 to 128 mL/min for females.
Time Frame: 18 months
Population: Data were not analyzed because the study was terminated early.
Groups:
- MMF, Prednisone: Induction Phase (Months 1 through 6): Participants received cyclophosphamide, 0.5 -1 g/m^2, IV once per month. Participants also received prednisone, 1 mg/kg/day, tablets (or methylprednisolone IV), PO; the dose was reduced by 5 mg every 2 weeks up to 20 mg/day, then reduced by 2.5 mg every 2 weeks to a final maintenance dose of 10 mg/day.
  Maintenance Phase (Months 7 through 12): Participants received MMF, 500 mg, tablets or capsules, PO, BID for 2 weeks; 500 mg, PO, TID for the next 2 weeks; 1 g, PO, BID for the remainder of the Maintenance Phase. Participants continued to receive maintenance prednisone (10 mg/day), as in the Induction Phase.
Arm/Group | MMF, Prednisone | Cyclophosphamide, Prednisone
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Urinary Protein
Description: Protein in urine is an indicator of kidney function. An increased urinary protein level indicates decreased kidney function. Normal values are approximately 0 to 8 milligrams per deciliter (mg/dL).
Time Frame: 18 months
Population: Data were not analyzed because the study was terminated early.
Arm/Group | MMF, Prednisone | Cyclophosphamide, Prednisone
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Serum Creatinine
Description: Serum creatinine is an indicator of kidney function. Creatinine is a substance formed from the metabolism of creatine, commonly found in blood, urine, and muscle tissue. It is removed from the blood by the kidneys and excreted in urine. An increased level of creatinine in the blood indicates decreased kidney function. Normal adult blood levels of creatinine are 0.5 to 1.1 mg/dL for females and 0.6 to 1.2 mg/dL for males, however the normal values are age-dependent as elderly participants typically have smaller muscle mass.
Time Frame: 18 months
Population: Data were not analyzed because the study was terminated early.
Arm/Group | MMF, Prednisone | Cyclophosphamide, Prednisone
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Serum Albumin
Description: Albumin is a protein made by the liver. A serum albumin test measures the amount of this protein in the clear liquid portion of the blood. Decreased serum albumin levels can be an indicator of liver and/or kidney disease, The normal range is 3.4 - 5.4 grams (g)/dL.
Time Frame: 18 months
Population: Data were not analyzed because the study was terminated early.
Arm/Group | MMF, Prednisone | Cyclophosphamide, Prednisone
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were reported starting with the first dose of study drug through the end of the study.
Description: The number of participants who were included and completed the study was very limited, so the data were not sufficient to be used for a statistical analysis to have a clinical results .
Arm/Group | MMF, Prednisone | Cyclophosphamide, Prednisone
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/6
Other Adverse Events (participants affected / at risk) | 0/5 | 2/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MMF, Prednisone (N=5) | Cyclophosphamide, Prednisone (N=6)
Cephalea (Nervous system disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2
Chills (General disorders) | 0 | 1
Swelling (General disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Data were not analyzed because the study was terminated early.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.